CLINICAL TRIAL: NCT07236307
Title: The Feasibility, Efficacy and Safety of UZit®: Single-arm Clinical Trial in Patients With Symptomatic Chronic Venous Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 244/CEFMUP/2024
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Venous Insufficiency of Leg; Drainage; Chronic Venous Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UZit® Intervention (Experimental)
  Interventions: Device: UZit®

INTERVENTIONS:
Device: UZit® — This is single-arm clinical trial to evaluate the effect of limb elevation with UZit®. Participants were invited to use UZit® overnight for one consecutive week to improve symptoms and signs of CVD of the lower limbs.
  UZit® (PPP-118717; technical Data Sheet in Supplementary Data 1) is an inflatable wedge-shaped device made of thermoplastic polyurethane (Figure 1), placed under a traditional mattress. When inflated, it creates an inclined plane of approximately 5%, optimizing venous circulation during rest. By evenly inclining the entire body, it avoids lumbar spine movement regardless of sleeping position.

SUMMARY:
The goal of this single-arm clinical trial is to learn whether overnight limb elevation using the UZit® device can improve symptoms and signs of chronic venous disease (CVD) in adults. The main questions it aims to answer are:

Does one week of overnight UZit® use improve quality of life in patients with CVD? Does UZit® use reduce ankle circumference and are there any adverse events associated with its use? Because there is no comparison group, all participants will use the UZit® device to determine whether these effects occur.

Participants will:

Use the UZit® device every night for one consecutive week. Follow their vascular surgeon's existing recommendations (e.g., compression stockings, venotonic medications).

Complete the CIVIQ-14 questionnaire at baseline and after one week of using the device to assess quality of life.

Measure ankle circumference twice daily (upon waking and before bedtime) using a digital tape measure, following marked anatomical points.

Report any symptoms-including low back pain-and rate their satisfaction with the device on a 0-5 scale.

DETAILED DESCRIPTION:
This single-arm clinical trial evaluates the effect of limb elevation with UZit®. Participants were invited to use UZit® overnight for one consecutive week to improve symptoms and signs of CVD of the lower limbs. UZit® (PPP-118717; technical Data Sheet in Supplementary Data 1) is an inflatable wedge-shaped device made of thermoplastic polyurethane (Figure 1), placed under a traditional mattress. When inflated, it creates an inclined plane of approximately 5%, optimizing venous circulation during rest. By evenly inclining the entire body, it avoids lumbar spine movement regardless of sleeping position. In addition to leg elevation, patients were advised to follow all other recommendations from their vascular surgeon (e.g., use of compression stockings, venotonic medications, etc.). The primary outcome was quality of life in CVD patients, assessed with the Portuguese translation of the CIVIQ-14 questionnaire, a validated and sensitive tool for detecting CVD-related changes. Patients completed the questionnaire at baseline and after one week of overnight UZit® use. Secondary outcomes included ankle circumference and adverse events. Ankle circumference was measured twice daily-immediately after waking and before bedtime-just above the malleolus, using a "Smart Tape Measure Body" digital device (resolution 0.1 cm, accuracy ±2%). Measurement points were marked on the skin with an "Edding 3000" marker, which patients refreshed daily. Participants were specifically asked about low back pain during limb elevation and any other symptoms during the intervention and the level of satisfaction using a scale from 0 to 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited from the outpatient setting of Casa de Saúde da Boavista, where they were evaluated due to worsening of their CVD symptoms

Exclusion Criteria:

* Peripheral artery disease
* Congestive heart failure
* Gastroesophageal reflux
* Inability to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Quality of life in CVD patients (CIVIQ-14 questionnaire) | One week of overnight UZit® use (baseline and after 1 week)
  CIVIQ (Chronic Venous Insufficiency Quality of Life Questionnaire); The score for each dimension was obtained by adding up the scores of each constituent item and the global index was obtained by adding up the scores of the items. Items were weighted equally. The minimum and maximum values of the scales are dependent on the number of items used in each of the dimensions and on the number of levels or categories for each item. In order to compare the mean scores between dimensions or scales, absolute scores were then converted into an index. For each dimension, we therefore obtained a result ranging from 0 to 100. In order to facilitate interpretation of the results, the scoring system can be reversed. According to this scoring method, improvement in quality of life between two study times is represented by an increase in score.

SECONDARY OUTCOMES:
Ankle circumference in CVD patients | One week without intervention (measurements taken twice daily) and one week with UZit® use (measurements taken twice daily)
Adverse events and participant satisfaction during UZit® use | One week of overnight UZit® use

CONTACTS AND LOCATIONS:
Locations (1):
- Casa da Saúde da Boavista, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided